CLINICAL TRIAL: NCT03533166
Title: Clinical and Microbiological Effects of a 0.03% Chlorhexidine Mouth Rinse in the Prevention of Peri-implant Diseases: a Randomized Clinical Trial
Brief Title: Effects of a 0.03% CHX Mouth Rinse in Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Dentaid SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15/064
Record Dates: First submitted 2018-04-18; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-implant mucositis; Chlorhexidine; CPC; Treatment
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Experimental): Mechanical treatment + 0.03% chlorhexidine + 0.05% CPC mouthrinse
  Interventions: Other: Chlorhexidine
- Placebo (Placebo Comparator): Mechanical treatment + Placebo mouth rinse
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Chlorhexidine — 0.03% Chlorhexidine + 0.05% CPC mouth rinse
  Arms: Chlorhexidine
Other: Placebo — Placebo mouth rinse
  Arms: Placebo

SUMMARY:
Aim: To evaluate the efficacy of a 0.03% chlorhexidine (CHX) and 0.05% cetyl pyridinium chloride (CPC) mouth rinse, as an adjunct to professionally and patient-administered mechanical plaque removal, in the treatment of peri-implant mucositis.

Material and Methods: Patients displaying peri-implant mucositis in, at least, one implant were included in this randomized, double-blinded, clinical trial. Subjects received a conventional professional prophylaxis (at baseline and 6-month visits) and were instructed to regular oral hygiene practices and to rinse, twice daily, during one year, with a 0.03% CHX and 0.05% CPC mouth rinse, or a placebo. Clinical, radiographic and microbiological data were recorded at baseline, 6 and 12 months. Disease resolution was defined as the absence of bleeding on probing (BOP). Repeated measures ANOVA, Student-t and chi square tests were used.

ELIGIBILITY:
Inclusion Criteria:

* the presence of, at least, one dental implant with clinical signs of peri-implant mucositis, defined as gently bleeding on probing (BOP) and/or suppuration without progressive radiographic bone loss (after at least 1 year of functional loading)

Exclusion Criteria:

* untreated or recurrent periodontitis [presence of nine or more sites with PD 5 mm and with full mouth bleeding score (FMBS) > 25%];
* implants affected by peri-implantitis, (BOP and/or suppuration and progressive radiographic bone loss);
* removable implant-retained prosthesis;
* history of intake of systemic antibiotics within the previous month or other chronic systemic medications that could interfere with the study outcomes;
* and women being pregnant or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Change on bleeding on probing on implants | Change baseline-12 months
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months. Primary outcome would be considered for the change between baseline and 12 months
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).

SECONDARY OUTCOMES:
Bleeding on probing (BOP) on implants | Baseline
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months.
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).
Bleeding on probing (BOP) on implants | 3 months
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months.
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).
Bleeding on probing (BOP) on implants | 6 months
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months.
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).
Bleeding on probing (BOP) on implants | 9 months
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months.
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).
Bleeding on probing (BOP) on implants | 12 months
  Bleeding on probing (BOP) on implants, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing (Jepsen et al. 2015) at baseline, 3, 6, 9 and 12 months.
  One blinded and calibrated investigator recorded BOP at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.78 for BOP).
Bleeding on probing (BOP) on teeth | Baseline
  Bleeding on probing (BOP) on teeth, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing
  One blinded and calibrated investigator recorded BOP at 6 sites around all teeth, using aPCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Bleeding on probing (BOP) on teeth | 6 months
  Bleeding on probing (BOP) on teeth, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing
  One blinded and calibrated investigator recorded BOP at 6 sites around all teeth, using aPCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Bleeding on probing (BOP) on teeth | 12 months
  Bleeding on probing (BOP) on teeth, evaluated dichotomously (presence/absence), considering a positive score when evident bleeding was observed within 15 s after gentle probing
  One blinded and calibrated investigator recorded BOP at 6 sites around all teeth, using aPCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Plaque on implants | Baseline
  Modified plaque index (MPlI) measured at six sites per implant (Mombelli et al. 1987):
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the implant;
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.79 for MPlI.
Plaque on implants | 6 months
  Modified plaque index (MPlI) measured at six sites per implant (Mombelli et al. 1987):
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the implant;
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.79 for MPlI.
Plaque on implants | 12 months
  Modified plaque index (MPlI) measured at six sites per implant (Mombelli et al. 1987):
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the implant;
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulting in kappa (k) values of 0.79 for MPlI.
Plaque on teeth | Baseline
  Modified plaque index (MPlI) measured at six sites per tooth
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the tooth
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Plaque on teeth | 6 months
  Modified plaque index (MPlI) measured at six sites per tooth
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the tooth
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Plaque on teeth | 12 months
  Modified plaque index (MPlI) measured at six sites per tooth
  * Score 0: no plaque detected;
  * Score 1: plaque only recognized by running the periodontal probe across the smooth marginal surface of the tooth
  * Score 2: plaque can be seen by the naked eye;
  * Score 3: abundance of soft matter.
  One blinded and calibrated investigator recorded MPI at 6 sites around teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Probing depth on implants | Baseline
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the peri-implant mucosal margin (six sites per implant).
  One blinded and calibrated investigator recorded PD at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient (ICC)=0.93 for PD.
Probing depth on implants | 6 months
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the peri-implant mucosal margin (six sites per implant).
  One blinded and calibrated investigator recorded PD at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient (ICC)=0.93 for PD.
Probing depth on implants | 12 months
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the peri-implant mucosal margin (six sites per implant).
  One blinded and calibrated investigator recorded PD at 6 sites around implants, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA)
  Calibration was achieved in double measurement calibration sessions, with a gold standard, on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient (ICC)=0.93 for PD.
Probing depth on teeth | Baseline
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the gingival margin (six sites per tooth).
  One blinded and calibrated investigator recorded PD at 6 sites around all teeth, using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Probing depth on teeth | 6 months
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the gingival margin (six sites per tooth).
  One blinded and calibrated investigator recorded PD at 6 sites around all teeth, using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Probing depth on teeth | 12 months
  Probing depth (PD) defined as the distance in mm, between the bottom of the pocket and the gingival margin (six sites per tooth).
  One blinded and calibrated investigator recorded PD at 6 sites around all teeth, using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Crown-length implant | Baseline
  Crown-length implant (CLI), defined as the distance in mm, between the incisal/occlusal portion of the crown and the peri-implant mucosal margin at the mid-buccal site.
  One blinded and calibrated investigator recorded CLI around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient of 0.96 for CLI.
Crown-length implant | 6 months
  Crown-length implant (CLI), defined as the distance in mm, between the incisal/occlusal portion of the crown and the peri-implant mucosal margin at the mid-buccal site.
  One blinded and calibrated investigator recorded CLI around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient of 0.96 for CLI.
Crown-length implant | 12 months
  Crown-length implant (CLI), defined as the distance in mm, between the incisal/occlusal portion of the crown and the peri-implant mucosal margin at the mid-buccal site.
  One blinded and calibrated investigator recorded CLI around the selected implant, using a plastic periodontal probe (PCV12, HuFriedy, Chicago, IL, USA).
  Calibration was achieved in double measurement calibration sessions, with a gold standard , on six randomly selected patients within one week. The inter-examiner agreement resulted in a intraclass correlation coefficient of 0.96 for CLI.
Recession on teeth | Baseline
  Recession (REC), defined as the distance in mm, between the gingival margin and the cements-enamel junction.
  One blinded and calibrated investigator recorded REC around all teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Recession on teeth | 6 months
  Recession (REC), defined as the distance in mm, between the gingival margin and the cements-enamel junction.
  One blinded and calibrated investigator recorded REC around all teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Recession on teeth | 12 months
  Recession (REC), defined as the distance in mm, between the gingival margin and the cements-enamel junction.
  One blinded and calibrated investigator recorded REC around all teeth using a PCP15 periodontal probe (HuFriedy® , Chicago, IL, USA).
Microbiological outcomes_total counts | Baseline
  Pooled subgingival samples were obtained from the two most inflamed accessible sites of the selected implant in each patient.
  Samples were taken with two consecutive sterile medium paper-points (#30, Maillefer, Ballaigues, Switzerland) that were kept in place for 10 s and then transferred into a screw-capped vial containing 1.5 ml of reduced transport fluid (RTF) (Syed & Loesche 1972). Samples were transported to the microbiology laboratory within 2 h, where aliquots of 0.1 mL were plated in different culture media.
  Counts were transformed in colony-forming units (CFU) per mL of the original sample. Total anaerobic counts and counts of selected periodontal pathogens (A. actinomycetemcomitans, Tannerella forsythia, Porphyromonas gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Eikenella corrodens, Campylobacter rectus and Fusobacterium nucleatum) were calculated.
Microbiological outcomes_total counts | 6 months
  Pooled subgingival samples were obtained from the two most inflamed accessible sites of the selected implant in each patient.
  Samples were taken with two consecutive sterile medium paper-points (#30, Maillefer, Ballaigues, Switzerland) that were kept in place for 10 s and then transferred into a screw-capped vial containing 1.5 ml of reduced transport fluid (RTF) (Syed & Loesche 1972). Samples were transported to the microbiology laboratory within 2 h, where aliquots of 0.1 mL were plated in different culture media.
  Counts were transformed in colony-forming units (CFU) per mL of the original sample. Total anaerobic counts and counts of selected periodontal pathogens (A. actinomycetemcomitans, Tannerella forsythia, Porphyromonas gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Eikenella corrodens, Campylobacter rectus and Fusobacterium nucleatum) were calculated.
Microbiological outcomes_total counts | 12 months
  Pooled subgingival samples were obtained from the two most inflamed accessible sites of the selected implant in each patient.
  Samples were taken with two consecutive sterile medium paper-points (#30, Maillefer, Ballaigues, Switzerland) that were kept in place for 10 s and then transferred into a screw-capped vial containing 1.5 ml of reduced transport fluid (RTF) (Syed & Loesche 1972). Samples were transported to the microbiology laboratory within 2 h, where aliquots of 0.1 mL were plated in different culture media.
  Counts were transformed in colony-forming units (CFU) per mL of the original sample. Total anaerobic counts and counts of selected periodontal pathogens (A. actinomycetemcomitans, Tannerella forsythia, Porphyromonas gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Eikenella corrodens, Campylobacter rectus and Fusobacterium nucleatum) were calculated.
Microbiological outcomes_frequency of detection | Baseline
  The frequency of detection was calculated as presence/absence of each periodontal pathogen
Microbiological outcomes_frequency of detection | 6 months
  The frequency of detection was calculated as presence/absence of each periodontal pathogen
Microbiological outcomes_frequency of detection | 12 months
  The frequency of detection was calculated as presence/absence of each periodontal pathogen
Microbiological outcomes_proportions | Baseline
  The proportions for each bacterial species was calculated by dividing the counts of each pathogen by the total counts.
Microbiological outcomes_proportions | 6 months
  The proportions for each bacterial species was calculated by dividing the counts of each pathogen by the total counts.
Microbiological outcomes_proportions | 12 months
  The proportions for each bacterial species was calculated by dividing the counts of each pathogen by the total counts.
Radiographic bone loss on implants | Baseline
  Standardized periapical radiographs using the parallel technique (Rinn® system, Dentsply, Weybridge, United Kingdom) were used to evaluate changes in the radiographic marginal bone levels (MBL).
  Scanned images were measured both at the mesial and distal sites using as landmarks the implant shoulder and the first bone implant contact (BIC) of the selected implant using an image analysis software (J-image).
  After a session of calibration (ICC=0.99), two investigators performed all the radiographic measurements.
Radiographic bone loss on implants | 3 months
  Standardized periapical radiographs using the parallel technique (Rinn® system, Dentsply, Weybridge, United Kingdom) were used to evaluate changes in the radiographic marginal bone levels (MBL).
  Scanned images were measured both at the mesial and distal sites using as landmarks the implant shoulder and the first bone implant contact (BIC) of the selected implant using an image analysis software (J-image).
  After a session of calibration (ICC=0.99), two investigators performed all the radiographic measurements.
Radiographic bone loss on implants | 12 months
  Standardized periapical radiographs using the parallel technique (Rinn® system, Dentsply, Weybridge, United Kingdom) were used to evaluate changes in the radiographic marginal bone levels (MBL).
  Scanned images were measured both at the mesial and distal sites using as landmarks the implant shoulder and the first bone implant contact (BIC) of the selected implant using an image analysis software (J-image).
  After a session of calibration (ICC=0.99), two investigators performed all the radiographic measurements.
Staining | Baseline
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Grundemann et al. 2000), recorded at nine areas per tooth (three mesial, three medial, three distal). Stain will be graded using the intensity stain index of Lobene (1968).
Staining | 6 months
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Grundemann et al. 2000), recorded at nine areas per tooth (three mesial, three medial, three distal). Stain will be graded using the intensity stain index of Lobene (1968).
Staining | 12 months
  Staining of teeth will be scored using the Gründemann modification of the stain index (GMSI) (Grundemann et al. 2000), recorded at nine areas per tooth (three mesial, three medial, three distal). Stain will be graded using the intensity stain index of Lobene (1968).
Adverse effect | Baseline
  A questionnaire will be filled to assess the patient-based variables and side effects, by the patients. They will be evaluated with a visual analogue scale (0-10)
Adverse effect | 6 months
  A questionnaire will be filled to assess the patient-based variables and side effects, by the patients. They will be evaluated with a visual analogue scale (0-10)
Adverse effect | 12 months
  A questionnaire will be filled to assess the patient-based variables and side effects, by the patients. They will be evaluated with a visual analogue scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Doctor, Principal Investigator — University Complutense Madrid (UCM); David Herrera, Doctor, Principal Investigator — University Complutense Madrid
Locations (1):
- Faculty of Dentistry, Univesity Complutense, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bollain J, Pulcini A, Sanz-Sanchez I, Figuero E, Alonso B, Sanz M, Herrera D. Efficacy of a 0.03% chlorhexidine and 0.05% cetylpyridinium chloride mouth rinse in reducing inflammation around the teeth and implants: a randomized clinical trial. Clin Oral Investig. 2021 Apr;25(4):1729-1741. doi: 10.1007/s00784-020-03474-3. Epub 2020 Jul 31. PMID 32737664
- [Derived] Pulcini A, Bollain J, Sanz-Sanchez I, Figuero E, Alonso B, Sanz M, Herrera D. Clinical effects of the adjunctive use of a 0.03% chlorhexidine and 0.05% cetylpyridinium chloride mouth rinse in the management of peri-implant diseases: A randomized clinical trial. J Clin Periodontol. 2019 Mar;46(3):342-353. doi: 10.1111/jcpe.13088. PMID 30779246